CLINICAL TRIAL: NCT03756415
Title: Evaluation of a New System to Clear CO2 During Noninvasive Ventilation (NIV)
Brief Title: CO2 Clearance During Noninvasive Ventilation (NIV)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Chief of Pulmonary and Critical Care, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Stefano Nava1
Record Dates: First submitted 2018-11-23; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Acute Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mask plus CO2 removal device (Experimental): a "traditional" mask with inserted a new CO2 removal device that is called DiMax Zero Total face mask "R",
  Interventions: Device: DiMax Zero Total face mask "R",
- traditional face mask (Active Comparator): Traditional mask without a CO2 clearance device inserted
  Interventions: Device: traditional face mask

INTERVENTIONS:
Device: DiMax Zero Total face mask "R", — a non-CO2 rebreathing device included directly in the full face mask
  Arms: mask plus CO2 removal device
Device: traditional face mask — a traditional mask without a non-CO2 rebreathing device included directly in the full face mask
  Arms: traditional face mask

SUMMARY:
In this randomized cross over study the investigators will evaluate the effects on gas exchange and patients' tolerance of a new CO2 non rebreathing devices incorporated in the mask vs the traditional mask COPD patients undergoing NIV for an episode of Acute Hypercapnia Respiratory Failure, will be randomized after at least 12 hour of ventilation to 1 h.trial with the usual full face mask or the same mask with the addition of a new CO2 clearance device

DETAILED DESCRIPTION:
In this randomized cross over study the investigators will evaluate the effects on gas exchange and patients' tolerance of a new CO2 non rebreathing devices incorporated in the mask vs the traditional mask COPD patients undergoing NIV for an episode of Acute Hypercapnia Respiratory Failure, will be randomized after at least 12 hour of ventilation to 1 h.trial with the usual full face mask (FM) or the same mask with the addition of a new CO2 clearance device (FM+d) In the interval between NIV sessions, arterial blood gases will be monitored and if PaCO2 will return to a baseline value with a tolerance of 10%, the patients will undergo another 1 h trial using the other mask.

The subjects will be studied in the sitting position and asked to relax throughout the period of the study.

The patients will be ventilated using pressure support ventilation (PSV) The order of use of the two interfaces will be determined for each patient by a previously generated randomized sequence.

FIO2 will be adjusted to obtain oxygen saturation around 92% at baseline and never modified throughout the study.

End-expiratory pressure will always fixed at 2 cm H2O, and trigger sensitivity will set at -0.5 cm H2O.

Inspiratory assistance during either PSV will be titrated to achieve a tidal volume between 6-8 mL/kg while avoiding occurrence of discomfort or visually assessed "wasted efforts".

The ventilatory settings will determined at the beginning of the first trial, and maintained unmodified throughout all the 3 runs.

Patient tolerance to NIMV, defined as the level of comfort using the different mask, will be assessed by means of a scale used and validated in previous studies that is defined as follows: 1, bad; 2, poor; 3, sufficient; 4, good; 5, very good. The patients were asked by the respiratory therapist to answer the following question: "How do the patient feel your breathing is using this mask?" The patient will give the score to the therapist at the end of each run, just before ABG measurements.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis
* sign inform consent
* able to tolerate the application of NIV

Exclusion Criteria:

* inability to tolerate the mask
* contraindication to NIV
* cancer, neurological diseases, and need of another life support besides the ventilator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
changes in arterial blood gases (ABGs) | immediate
  Recording of carbon dioxide arterial tensione and oxygen arterial tension using an arterial puncture performed in the radial artery
patient's tolerance to the mask | immediate
  the tolerance will be recorded using an ad hoc scale

CONTACTS AND LOCATIONS:
Overall Officials: stefano nava, Principal Investigator — Azienda Ospedaliera Sant'Orsola

IPD SHARING:
Plan to Share IPD: No
not allow to release individual data